CLINICAL TRIAL: NCT01739491
Title: A Post-Marketing Surveillance Study on the Safety And Effectiveness of Bendamustine Hydrochloride Among Adult Filipino Patients With Chronic Lymphocytic Leukemia
Brief Title: A Study of Safety and Effectiveness of Bendamustine Hydrochloride in Adult Filipino Patients With Chronic Lymphocytic Leukemia
Status: Withdrawn | Type: Observational
Why Stopped: The study is cancelled. FDA Circular 2013-004 mandates that PMSs like this are not required
Sponsor: Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100917; BENDAMUSCLL4001 (Other: Jannsen Pharmaceutica)
Record Dates: First submitted 2012-11-29; First posted 2012-12-03 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic lymphocytic leukemia; Bendamustine hydrochloride; Leukemia; Filipino
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bendamustine hydrochloride: Adult Filipino patients with chronic lymphocytic leukemia will be taking bendamustine hydrochloride as per the dosing regimen given on product insert approved in Philippines.
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — This is an obeservational study. Bendamustine hydrochloride will be administered (as per product insert) through intravenous infusion over 30-60 minutes at 100 mg/meter square body surface area on days 1 and 2 of a 28-day cycle.

SUMMARY:
The purpose of this study is to assess safety and effectiveness of extended bendamustine in the treatment of chronic lymphocytic leukemia (CLL).

DETAILED DESCRIPTION:
This is a Phase IV, open label (all people know the identity of the intervention), multi-center, observational (a scientific study to make a clear and easy understanding of the cause and effect relationship) study of bendamustine. The study duration is of 24 Weeks to coincide with the 4 weeks-6 cycles bendamustine treatment. The study will run for three years, and will enroll 10 percent of patient who would use this product, as a requirement of the Philippine Food and Drug Administration (FDA). Approximately fifty patients will be enrolled in this study. Safety evaluations including adverse events, clinical laboratory tests, electrocardiogram, vital signs, and physical examination will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult Filipino patients with chronic lymphocytic leukemia
* Patients who are cytologically-diagnosed with chronic lymphocytic leukaemia (symptomatic Binet stage B or C) and for whom fludarabine combination chemotherapy is not appropriate
* World health organization performance Status of 0, 1, or 2
* Need-to-treat criteria in B-cell chronic lymphocytic leukemia

Exclusion Criteria:

* Had received previous treatment with other cytotoxic drugs
* Had a history of a second malignancy (except cured basal cell carcinoma or cured cervical cancer)
* Concomitant illnesses such as overt heart failure, cardiomyopathy, myocardial infarction within the last 6 months, severe uncontrolled diabetes mellitus, severe uncontrolled hypertension, active infection that required systemic antibiotic treatment in an investigational drug study within 30 days prior to selection
* Patients with severe renal and hepatic impairment
* Patients with severe bone marrow suppression and severe blood count alterations
* Pregnant women and lactating mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult Filipino patients who are diagnosed with chronic lymphocytic leukemia.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients with incidence of adverse events | Up to Week 24
Number of patients with incidence of discontinuation of study medication due to adverse events | Up to Week 24

SECONDARY OUTCOMES:
Number of patients who show complete remission | Week 4, Week 8, Week 12, Week 16, Week 20, Week 24
  Number of patients with complete remission will be evaluated using the National Cancer Institute-Sponsored Working Group (NCISWG) criteria.
Number of patients who show partial remission | Week 4, Week 8, Week 12, Week 16, Week 20, Week 24
  Number of patients with partial remission will be evaluated using the National Cancer Institute-Sponsored Working Group (NCISWG) criteria.
Number of patients with stable disease | Week 4, Week 8, Week 12, Week 16, Week 20, Week 24
  Number of patients with stable disease will be evaluated using the National Cancer Institute-Sponsored Working Group (NCISWG) criteria.
Number of patients who show disease progression | Week 4, Week 8, Week 12, Week 16, Week 20, Week 24
  Number of patients with disease progression will be evaluated using the National Cancer Institute-Sponsored Working Group (NCISWG) criteria.
Number of patients with lack of effect (failure of expected pharmacologic action) | Week 4, Week 8, Week 12, Week 16, Week 20, Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Jannsen Pharmaceutica Clinical trial, Study Director — Jannsen Pharmaceutica